CLINICAL TRIAL: NCT02556255
Title: Safety and Effectiveness Evaluation of Eximo's B-Laser™ Atherectomy Device, in Subjects Affected With PAD
Brief Title: Safety and Effectiveness Study of Eximo's B-Laser™ Atherectomy Device for PAD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eximo Medical Ltd. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EX-PAD-01
Record Dates: First submitted 2015-09-02; First posted 2015-09-22 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Peripheral Artery Disease; PAD; Atherosclerosis; Arterial Occlusive Diseases; Peripheral Vascular Diseases; PVD
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis; Arterial Occlusive Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- B-Laser™ Atherectomy Catheter (Experimental): Percutaneous Transluminal Angioplasty (PTA) for treatment of infrainguinal arteries in patients with Peripheral Artery Disease (PAD), that the atherectomy part of the PTA will include an experimental atherectomy catheter, B-Laser™.
  Interventions: Device: B-Laser™ Atherectomy Catheter

INTERVENTIONS:
Device: B-Laser™ Atherectomy Catheter — Laser atherectomy catheter based on 355 nm

SUMMARY:
The aim of the study is to assess the safety and efficacy of the use of the Eximo's B-Laser™ catheter in subjects affected with Peripheral Artery Disease (PAD) in lower extremity arteries.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, international, open-label, non-randomized clinical study.

All enrolled subjects will undergo atherectomy procedure, during which the B-Laser™ catheter will be used to perform atherectomy in target lesion, followed by any other adjunctive therapy (balloon and/or stent etc.). The procedure will be done according to standard hospital procedure for atherectomy. The steps of the operation before and after the operating of the B-Laser™ device are routinely used practice and will be done according to local practice at each hospital. For the post-atherectomy stage, as an adjunctive therapy in the procedure, any approved device may be used (balloon and/or stent etc.).

Subjects will then be followed for 12 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old.
2. Subject is a candidate for endovascular intervention for peripheral artery disease in the lower extremities.
3. Documented symptomatic atherosclerotic peripheral artery disease Rutherford Classification 2-4.
4. Subject has infrainguinal target lesion(s) with any type of stenosis (naïve or recurrent) estimated to be ≥70% based on CT angiogram or other imaging modality.
5. At least one patent tibial run-off vessel at baseline.
6. Subject is capable and willing to comply with the scheduled follow up.
7. Subject is able and willing to sign a written informed consent form (ICF).

Intraoperative inclusion criteria (by fluoroscopy angiogram):

1. Reference vessel lumen diameter proximal to target lesion is ≥150% of the outer diameter of the B-Laser™ to be used.
2. Target lesion has been crossed with a guidewire within the true lumen.
3. Target lesion has a stenosis estimated to be ≥70%.

Exclusion Criteria:

1. Target lesion is in a vessel graft or synthetic graft.
2. Target lesion length >25 cm.
3. Endovascular or surgical procedure performed less than or equal to 30 days prior to the index procedure OR Planned endovascular or surgical procedure 30 days after the index procedure.
4. Intent to use other atherectomy device in the same procedure.
5. Flow limiting dissection proximal to, distal to or in the target lesion.
6. Evidence or history of intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stroke within the past 2 months.
7. Evidence or history of aneurysm in the target vessel within the past 2 months.
8. History of bleeding diathesis, coagulopathy or inability to accept blood transfusions.
9. History of heparin-induced thrombocytopenia (HIT).
10. Significant acute or chronic kidney disease with a creatinine level >2.5 mg/dl, and/or requiring dialysis.
11. Any thrombolytic therapy within 2 weeks of the index procedure.
12. History of severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days.
13. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
14. Subjects in whom anti-platelet, anticoagulant, or thrombolytic therapy is contraindicated.
15. Serious illness that may affect subject compliance to protocol and at a minimum the 30-day follow-up.
16. Participating in other clinical study that involves any kind of intervention, including pharmaceutical.
17. Issue that in the judgment of the investigator, may affect the results of the study.
18. Subject is pregnant or planning to become pregnant during the study period.

Intraoperative exclusion criteria (by fluoroscopy angiogram):

1. Total occlusion of the Target lesion that cannot be crossed in the true lumen by 0.014" GW.
2. Target lesion length >25 cm.
3. Reference vessel lumen diameter proximal to target lesion is <150% of the outer diameter of the B-Laser™.
4. Any clinical and/or angiographic complication attributed to the use of another device prior to the study procedure.
5. Flow limiting dissection proximal, distal or in the target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oshrat Cohen, Ph.D., MBA, Study Director — Angiodynamics, Inc.; Waclaw Kuczmik, Dr., Principal Investigator — Górnośląskie Centrum Medyczne im. prof. Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach; Grzegorz Oszkinis, Prof., Principal Investigator — Poznan Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im.Karola Marcinkowskiego; Lukasz Dzieciuchowicz, Prof, Principal Investigator — Poznan Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im.Karola Marcinkowskiego; Lukasz Kruszyna, Prof, Principal Investigator — Poznan Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im.Karola Marcinkowskiego
Locations (2):
- Poland (2):
  - Gornoslaskie Centrum Medyczne im. prof. Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan

RESULTS

PARTICIPANT FLOW:
Groups:
- B-Laser™ Atherectomy Catheter: Percutaneous Transluminal Angioplasty (PTA) for treatment of infrainguinal arteries in patients with Peripheral Artery Disease (PAD) that the atherectomy part of the PTA includes an experimental atherectomy catheter, B-Laser™.
Period: Overall Study
Arm/Group | B-Laser™ Atherectomy Catheter
Started | 50
Completed | 46
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ABI (Ankle Brachial Index) [Mean (Standard Deviation); unit: ratio] — ABI is calculated as the ratio of the ankle blood pressure to the arm blood pressure. The normal value ranges between 0.9 to 1.3. Higher ABI score represents a better outcome
  ratio | 0.57 (0.14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 30 Day Freedom From Major Adverse Events
Description: 1. Need for emergency surgical revascularization of the target limb
  2. Unplanned target limb amputation above the ankle
  3. Clinically driven Target Lesion Revascularization (TLR)
  4. Cardiovascular related deaths
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Participants | 50

2. Primary Outcome: Number of Participants With Perioperative (Until Discharge) Freedom From Device/Procedure* Related Adverse Events (1)
Description: (*NOTE: Device- or procedure-related AE refers only to the ATHERECTOMY PROCEDURE (with B-Laser™) and not the entire index procedure.)
  1. Clinically Significant Perforations requiring intervention
  2. Clinically Significant Dissections requiring intervention
  3. Clinically Significant Embolus requiring intervention
  4. Clinically Pseudo-aneurysm requiring intervention
Time Frame: Perioperative (until discharge), an average of 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Participants | 50

3. Primary Outcome: Number of Lesions With Technical Success Rate: the Ability of the B-Laser™ Catheter to Cross the Target Lesion Stenosis Over the Wire.
Description: The technical success will be evaluated visually by the performing physician during procedure by fluoroscopy. It is evaluated per lesion and not per subject
Time Frame: Intraoperative (during the index procedure, after B-Laser™ catheter crossing, before adjunctive therapy)
Population: Generally angiographic outcomes are evaluated per lesions (53) and not per participants (50). Yet, this specific endpoint is analyzed for 52 lesions (instead of 53), since the data for this timepoint in one participant with one lesion was missing for evaluation of this specific endpoint.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 49
Number analyzed (lesions) | 52
lesions | 52

4. Secondary Outcome: Number of Participants With Perioperative (Until Discharge) Freedom From Device/Procedure* Related Adverse Events (2)
Description: (*NOTE: Device- or Procedure-related AE Refers Only to the ATHERECTOMY PROCEDURE (With B-Laser™) and Not the Entire Index Procedure.)
  1. Emboli, defined as a new occlusion of any visualized runoff vessel which cannot be reversed with an intravascular vasodilator
  2. Flow limiting dissection
Time Frame: Perioperative (until discharge), an average of 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Participants | 50

5. Secondary Outcome: Number of Participants With 30 Day Freedom From Device/Procedure* Related Adverse Events
Description: (*NOTE: Device- or Procedure-related AE Refers Only to the ATHERECTOMY PROCEDURE (With B-Laser™) and Not the Entire Index Procedure.)
  1. Clinically Significant Dissections requiring intervention
  2. Clinically Significant Embolus requiring intervention
  3. Clinically Pseudo-aneurysm requiring intervention
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Participants | 50

6. Secondary Outcome: Number of Lesions With Post-intervention Residual Diameter Stenosis of <30% With Adjunctive Therapy Assessed by Fluoroscopic Angiography in Cases Where Adjunctive Therapy is Medically Applicable
Description: The ability of the B-Laser™ catheter to achieve a post-intervention residual diameter stenosis of <30% with adjunctive therapy assessed by fluoroscopic angiography in cases where adjunctive therapy is medically applicable
Time Frame: Intraoperative (at the end of the index procedure, after the last adjunctive therapy, e.g. last balloon or last stent)
Population: This endpoint is analyzed for lesions (53) and not for participants (50)
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Number analyzed (lesions) | 53
lesions | 38

7. Secondary Outcome: Change in Ankle-Brachial Index (ABI) Post B-Laser™ Device Procedure Compared to Baseline
Description: Change in Ankle-Brachial Index (ABI) post B-Laser™ device procedure compared to baseline.
  ABI is calculated as the ratio of the ankle blood pressure to the arm blood pressure. The normal value ranges between 0.9 to 1.3.
  The change is calculated as the value at the later time point minus the value at the earlier time point, when positive results represent increases while negative results represent decrease, so higher ABI score at the later time point represents an improvement through time and vice versa.
Time Frame: baseline and 30 days, 6 months and 12 months post procedure
Population: The number analyzed in one or more rows differs from overall number since it excludes missing data at different time-points
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
ratio
  baseline | 0.57 (0.14)
  30 days | 0.94 (0.14)
  6 months: number analyzed (Participants) | 48
  6 months | 0.84 (0.20)
  12 months: number analyzed (Participants) | 29
  12 months | 0.77 (0.16)

8. Secondary Outcome: Change in Rutherford Classification Post B-Laser™ Device Procedure Compared to Baseline
Description: Change in Rutherford Classification Post B-Laser™ Device Procedure Compared to Baseline.
  Rutherford Classification has seven stages, from Stage 0 to Stage 6, when the lower value indicate a better outcome: 0= Asymptomatic; 1= Mild claudication; 2= Moderate claudication; 3= Severe claudication; 4= Rest pain; 5= Ischemic ulceration not exceeding ulcer of the digits of the foot; 6= Severe ischemic ulcers or frank gangrene.
  The change is calculated as the value at the later time point minus the value at the earlier time point, when positive results represent decrease while negative results represent increases, so lower Rutherford score at the later time point represents an improvement through time and vice versa.
Time Frame: baseline and 30 days, 6 months and 12 months post procedure
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Participants
  baseline: Rutherford class 0 | 0
  baseline: Rutherford class 1 | 0
  baseline: Rutherford class 2 | 10
  baseline: Rutherford class 3 | 35
  baseline: Rutherford class 4 | 5
  30 days: Rutherford class 0 | 24
  30 days: Rutherford class 1 | 21
  30 days: Rutherford class 2 | 3
  30 days: Rutherford class 3 | 2
  30 days: Rutherford class 4 | 0
  6 months: number analyzed (Participants) | 48
  6 months: Rutherford class 0 | 23
  6 months: Rutherford class 1 | 12
  6 months: Rutherford class 2 | 8
  6 months: Rutherford class 3 | 5
  6 months: Rutherford class 4 | 0
  12 months: number analyzed (Participants) | 29
  12 months: Rutherford class 0 | 8
  12 months: Rutherford class 1 | 11
  12 months: Rutherford class 2 | 6
  12 months: Rutherford class 3 | 4
  12 months: Rutherford class 4 | 0

9. Secondary Outcome: Change in Grade of Walking Impairment Questionnaire (WIQ) Post B-Laser™ Device Procedure Compared to Baseline
Description: Change in Grade of Walking Impairment Questionnaire (WIQ) Post B-Laser™ Device Procedure Compared to Baseline. WIQ score ranges from 0-100 with higher score indicating a better walking outcomes.
  The change is calculated as the value at the later time point minus the value at the earlier time point, when positive results represent increases while negative results represent decrease, so higher WIQ score at the later time point represents an improvement through time and vice versa.
Time Frame: baseline and 30 days, 6 months and 12 months post procedure
Population: The number analyzed in one or more rows differs from overall number since it excludes missing data at different time-points.
  Answers to all questions in the Walking Impairment Questionnaire (WIQ) must be provided to obtain a valid result, incomplete questionnaires were not considered.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 49
score on a scale
  baseline | 34.16 (8.15)
  30 days | 71.72 (19.88)
  6 months: number analyzed (Participants) | 45
  6 months | 67.84 (22.05)
  12 months: number analyzed (Participants) | 21
  12 months | 53.30 (18.09)

10. Post Hoc Outcome: Number of Lesions With Post-intervention Residual Diameter Stenosis of ≤30% With Adjunctive Therapy Assessed by Fluoroscopic Angiography in Cases Where Adjunctive Therapy is Medically Applicable
Description: EX-PAD-01 study secondary efficacy endpoint of the post adjunctive therapy residual diameter stenosis, was set per protocol with a threshold at <30%, however, in many other atherectomy studies, this threshold is set at ≤30%, Therefore results with this threshold are presented as well
Time Frame: Intraoperative (at the end of the index procedure, after the last adjunctive therapy, e.g. last balloon or last stent)
Population: This endpoint is analyzed for lesions (53) and not for participants (50)
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | B-Laser™ Atherectomy Catheter
Number analyzed (Participants) | 50
Number analyzed (lesions) | 53
lesions | 48

ADVERSE EVENTS:
Time Frame: 30 days, 6 months and 12 months post procedure with B-Laser™ device
Description: If multiple terms (events) were coded within 1 reported event in eCRF, they were connected with '@' sign. E.g. LLT terms 'Upper gastrointestinal hemorrhage@Esophagitis@Gastroesophageal reflux disease' denotes the event description reported in eCRF: 'Upper gastrointestinal hemorrhage (mild) occurred on 15.03, resulted in hospitalization between 28-31.03. During hospital stay chest CT was done and endoscopic evaluation of upper GI tract, that revealed esophagitis, gastroesophageal reflux disease'.
Arm/Group | B-Laser™ Atherectomy Catheter
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 14/46
Other Adverse Events (participants affected / at risk) | 15/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-Laser™ Atherectomy Catheter (N=46)
Angina Pectoris (Cardiac disorders) | 1 (1) — 329 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Heart Failure (Cardiac disorders) | 2 (2) — 144 & 356 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Chronic ischemic heart disease, unspecified (Cardiac disorders) | 1 (1) — 82 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Non STEMI@Atrioventricular block@Cardiogenic shock@Acute renal failure (Cardiac disorders) | 1 (1) — 322 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) — 8 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Large intestine angiodysplasia (Gastrointestinal disorders) | 1 (1) — 126 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Upper gastrointestinal hemorrhage@ Esophagitis@ Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — 92 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Vascular access site hematoma (Injury, poisoning and procedural complications) | 2 (2) — 0 days post procedure. Not related to the Investigational Device. Causal relationship to the index procedure.
Superficial femoral arterial stenosis & Claudication@Leg ischemia@Disease progression (Vascular disorders) | 2 (2) — 8 & 197 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Leg ischemia@Superficial femoral arterial stenosis@Claudication (Vascular disorders) | 1 (1) — 384 days post procedure. Not related to the Investigational Device. Possibly related to the index procedure.
Non STEMI@ Bradycardia (Cardiac disorders) | 1 (1) — 319 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Angina pectoris unstable (Cardiac disorders) | 1 (1) — 308 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Atrial fibrillation (Cardiac disorders) | 1 (1) — 319 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Leg ischemia@ Popliteal arterial restenosis (Vascular disorders) | 1 (1) — 245 days post procedure. Might be related to both device or Index procedure and judged to be more due to Index procedure.
Intracranial hemorrhage (Nervous system disorders) | 1 (1) — 232 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-Laser™ Atherectomy Catheter (N=46)
Vascular dissection (Vascular disorders) | 3 (3) — 0 days post procedure. Not related to the Investigational Device. Definitely related to the index procedure. Minor dissection.
Arterial occlusion (Vascular disorders) | 1 (1) — 163 days post procedure. Not related to the Investigational Device. Related to the index procedure.
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — 0 days post procedure. Not related to the Investigational Device. Definitely related to the index procedure.
Leg ischemia@Superficial femoral arterial stenosis (Vascular disorders) | 4 (4) — 195 & 207 & 221 & 324 days post procedures. Not related to the Investigational Device. Probably not related to the index procedure.
Leg ischemia (Vascular disorders) | 1 (1) — 188 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Claudication (Vascular disorders) | 1 (1) — 31 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Nasal bleeding (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 20 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — 287 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Skin infection (Infections and infestations) | 1 (1) — 180 days post procedure. Not related to the Investigational Device. Not related to the index procedure.
Edema lower limb (General disorders) | 2 (2) — 4 & 28 days post procedure. Not related to the Investigational Device. Not related to the index procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02556255/Prot_SAP_000.pdf